CLINICAL TRIAL: NCT05965713
Title: IpsiHand Device Use in Hemiparetic Stroke Population to Assess Home Based EEG System Candidacy for BCI Rehabilitation of the Upper Extremity and the Efficacy of a Full Remote Home Based BCI Therapy - A Randomized Control Trial
Brief Title: National Fully Remote Use of IpsiHand Device in Hemiparetic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolutions, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: National Remote IpsiHand Study; 4R44HD105579-02 (NIH)
Record Dates: First submitted 2023-07-18; First posted 2023-07-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Hemiparesis; Spasticity as Sequela of Stroke; Brain Computer Interface
Keywords: Neurolutions; IpsiHand
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Study staff will screen participants virtually or in person for eligibility after completing the informed consent process and documentation. After screening for study eligibility has occurred, the initial EEG screening will take place for all individuals who meet the criteria for the study as to ensure no preference to subjects with optimal signals for use of the IpsiHand. Once EEG screenings have been completed, the participant will be randomly assigned to Group 1 (BCI treatment) or Group 2 (standard of care treatment group). Each group will complete a daily therapy regimen. In Group 1 (BCI group)- will complete daily BCI therapy. In Group 2 (standard of care)- individuals will complete standard of care therapy program daily for 12 weeks provided by an occupational therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BCI treatment Group using the IpsiHand (Experimental): Phase 1: Group 1 subjects will receive an IpsiHand Screening System to complete a remote EEG Screening. Subjects will undergo an EEG screening protocol to ensure that a consistent control signal will be present to control the IpsiHand device. After an EEG screening session is complete, the participants screening data will be analyzed to ensure that sufficient cortical signals are present. Randomization for assignment to group 1 or 2 will then occur. Once assigned to group 1, if consistent signals are found, the participant will then continue to Phase 2.
  Phase 2: Group 1 subjects will be provided with a Neurolutions IpsiHand BCI system, which combines a novel powered exoskeleton with a commercial EEG amplifier and active electrode system. The exoskeleton opens and closes the patient's hand in a three-finger pinch grip. Patients will use the BCI system on a minimum of 5 days per week for 12 weeks. Patients will complete five or more 10-minute runs of the BCI task per day.
  Interventions: Device: Neurolutions IpsiHand System
- Standard of Care - Home Exercise Program for Upper Extremity (Experimental): Phase 1: Group 1 subjects will receive an IpsiHand Screening System to complete a remote EEG Screening. Once randomized, the participant will be assigned to group 2 to begin standard of care treatment at home.
  Phase 2: After being assigned to Group 2, subjects will serve as the control group in the study. Subjects will receive a customized home range of motion exercise program. Subjects will be recommended to complete their exercises daily, 5 out of 7 days per week for 12 weeks to control for the non-specific motor and sensory effects of BCI training. To help ensure compliance with the at-home portion of the protocol in the control group, participants will receive daily virtual monitoring from the study clinical specialist.
  Interventions: Other: Standard of Care - Home Exercise Program for Upper Extremity

INTERVENTIONS:
Device: Neurolutions IpsiHand System — The IpsiHand system utilizes a Brain-Computer Interface (BCI) to enable operation of a robotic hand exoskeleton worn on the hand and wrist as participants are guided through a rehabilitation program on a tablet. Participants will complete 12 weeks of home therapy with the IpsiHand system. Motor function of their impaired upper extremity will be evaluated at baseline and at 12 weeks completion of IpsiHand use.
  Arms: BCI treatment Group using the IpsiHand
Other: Standard of Care - Home Exercise Program for Upper Extremity — Subjects will receive a customized standard of care home exercise program. Subjects will be recommended to complete their exercises daily, 5 out of 7 days per week for 12 weeks.
  Arms: Standard of Care - Home Exercise Program for Upper Extremity

SUMMARY:
The goal of this study is to define the efficacy of fully remote home-based BCI therapy in chronic hemiparetic subcortical stroke patients. A randomized controlled study using the integrated remote BCI system will be tested against standard exercise therapy to determine the efficacy of motor improvement in chronic stroke patients with an upper extremity hemiparesis. Specifically, the integrated BCI system will include 1) the remote screening and motor assessment system for the upper extremity and 2) the BCI-controlled robotic hand exoskeleton (i.e. IpsiHand).

DETAILED DESCRIPTION:
The ultimate goal of this project is to develop a functioning and clinically feasible method for restoring function to motor impaired stroke survivors. This ultimate goal is to develop a system that allows for enhanced functional capability and works consistently over a long-term basis and is accessible remotely no matter location or access to healthcare. In developing a new rehabilitation method, the researchers hope to create a system that allows for closed loop feedback through a robotic hand orthosis on the motor impaired side of stroke patients in response to intended movements of the muscles. The method, if successful, would represent an ideal, non-invasive method of promoting motor learning and recovery in stroke survivors. The ability to operate robotic hand orthosis using electrical signals of the brain is rapidly leaving the realm of science fiction and becoming a realistic goal of the clinical community. The current advances in BCI controlled neuroprosthetics could have immeasurable influence on adult patients with severe motor impairments from stroke. Even further on the horizon the insights developed from such work could substantively alter the way all stroke patients are treated and rehabilitated.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age (18-85)
2. Adults who sustained a CVA
3. Have upper extremity hemiparesis/hemiplegia
4. Participants who are not receiving Botox Injections for the upper extremity may be included. Should a participant be receiving Botox injections for the upper extremity, they may be included but Botox administration must be timed to coincide within a week of the beginning of training.

Exclusion Criteria:

1. Participants who are not receiving Botox Injections for the upper extremity may be included. Should a participant be receiving Botox injections for the upper extremity, they may be included but Botox administration must be timed to coincide within a week of the beginning of training.
2. Participants who are too cognitively impaired to understand the task or provide informed consent will be excluded. A Short-Blessed Test score of 8 or more will be excluded.
3. Participants who have contractures in the affected wrist and digits will be excluded, as the device will not comfortably fit.
4. Participants who have receptive aphasia and unable to follow written directions will be excluded. A score of 6 or less on the MS Aphasia Screening Test will be excluded.
5. Participants receiving any formal upper extremity therapy will be excluded.
6. Participants with ataxia apraxia or severe psychiatric illness (other than post stroke depression) will be excluded.
7. Participants who are pregnant or breast-feeding will be excluded.
8. Participants who have nerve or sensory impairment that may limit or interfere with their ability to sense pain will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer - Upper Extremity (UEFM) , Manual Long Form | Assessed at baseline visit and at completion of study
  Valid assessment tool of upper extremity motor function in persons chronic stroke with moderate to severe deficits. Lowest score 0, highest score 66.

SECONDARY OUTCOMES:
Neurolutions Upper Extremity Remote Assessment (Remote Digital Fugl Meyer) | Baseline, 2 week, 4 week, 6 week, 8 week, 10 week and 12 week completion assessment
  Shortened and validated digitized assessment tool derived from the Fugl-Meyer Long form developed by Neurolutions of upper extremity motor function in persons chronic stroke with moderate to severe deficits. Embedded into study software. Lowest score 0, highest score 66.
Pinch force (Dynamometer) | Baseline and 12 week completion assessment
  Evaluation of two and three point pinch strength via dynamometry; lowest score= 0lbs, highest score =150lbs
Gross Grasp (Dynamometer) | Baseline and 12 week completion assessment
  Evaluation of gross grasp strength via dynamometry; lowest score= 0lbs, highest score =150lbs
Motricity Index (Shoulder, Elbow, Pinch) | Baseline and 12 week completion assessment
  Evaluation of motor strength on the shoulder, elbow and pinch. Scored on a 0-5 scale. 0 being totally absent muscle strength and range of motion, 5 bring full strength and range of motion of limb.
Western Aphasia Battery (Bedside Record Form) | Baseline and 12 week completion assessment
  Assessment of language function for classification of aphasia following a stoke.
Timed Up and Go Test (TUG) | Baseline and 12 week completion assessment
  Assessment functional mobility and fall risk
10 Meter Walking Test | Baseline and 12 week completion assessment
  Assessment functional mobility, speed of mobility and fall risk
Arm Motor Ability Test (4 Subtests Only) | Baseline and 12 week completion assessment
  Assessment to evaluate upper extremity function in activities of daily living
Trail Making Test- Parts A and B | Baseline and 12 week completion assessment
  Assessment of general cognitive function specifically assesses working memory, visual processing, visuospatial skills, selective and divided attention.
Modified Rankin Scale | Baseline and 12 week completion assessment
  A widely used assessment tool for measuring the degree of disability or dependence in people who have experienced stroke or other neurological conditions. The sale ranges from 0 (no symptoms) to 6 (death), and is commonly used as a primary outcome measure in stroke clinical trials.
PHQ-9 | Baseline and 12 week completion assessment
  A widely used assessment tool for self reporting of depression. This assessment is scored from 0-27.
  0-4: Minimal or no depression. 5-9: Mild depression. 10-14: Moderate depression. 15-19: Moderately severe depression. 20-27: Severe depression.
Zarit Burden Interview (ZBI) | Baseline and 12 week completion assessment
  Widely used questionnaire designed to assess the level of burden experienced by caregivers
The Barthel Index | Baseline and 12 week completion assessment
  Assessment tool that measures a person's functional independence in activities of daily living and self-care

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Carter, MD, PhD, Principal Investigator — Washington University in Saint Louis
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A variables associated with occupational and physical therapy stroke rehabilitation utilization and outcomes — https://pubmed.ncbi.nlm.nih.gov/15839599/
- See also: Inequities in access to inpatient rehabilitation after stroke: an international scoping review — https://pubmed.ncbi.nlm.nih.gov/28835194/
- See also: Clinical practice. Rehabilitation after stroke — https://pubmed.ncbi.nlm.nih.gov/15843670/
- See also: Brain-Computer Interface in Stroke Rehabilitation — http://koreascience.or.kr/article/JAKO201319133640292.page
- See also: Think to move: a neuromagnetic brain-computer interface (BCI) system for chronic stroke — https://pubmed.ncbi.nlm.nih.gov/18258825/
- See also: Feasibility of a new application of noninvasive Brain Computer Interface (BCI): a case study of training for recovery of volitional motor control after stroke — https://pubmed.ncbi.nlm.nih.gov/20208465/
- See also: Brain-computer interface-based robotic end effector system for wrist and hand rehabilitation: results of a three-armed randomized controlled trial for chronic stroke — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4114185/
- See also: An evaluation framework for a rural home-based telerehabilitation network — https://pubmed.ncbi.nlm.nih.gov/16235812/
- See also: Disparities in postacute stroke rehabilitation disposition to acute inpatient rehabilitation vs. home: findings from the North Carolina Hospital Discharge Database — https://pubmed.ncbi.nlm.nih.gov/19169175/
- See also: Barriers to care among racial/ethnic groups under managed care — https://pubmed.ncbi.nlm.nih.gov/10916961/
- See also: Stroke patients' and carers' perception of barriers to accessing stroke information — https://pubmed.ncbi.nlm.nih.gov/20542850/
- See also: Rehabilitation with poststroke motor recovery: a review with a focus on neural plasticity — https://pubmed.ncbi.nlm.nih.gov/23738231/
- See also: Brain-computer interface with somatosensory feedback improves functional recovery from severe hemiplegia due to chronic stroke — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4083225/
- See also: Efficacy of brain-computer interface-driven neuromuscular electrical stimulation for chronic paresis after stroke — https://pubmed.ncbi.nlm.nih.gov/24590225/